CLINICAL TRIAL: NCT06010628
Title: Intravenous Tenecteplase for Acute Ischemic Stroke Within 4.5 to 6 Hours of Onset (EXIT-BT2): a Prospective, Randomized, Open Label, Blinded Endpoint, and Multi-center Study
Brief Title: Tenecteplase for Acute Ischemic Stroke Within 4.5 to 6 Hours of Onset (EXIT-BT2)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2023) 144
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Ischemic
Keywords: thrombolysis
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase group (Experimental): intravenous thrombolysis with tenecteplase
  Interventions: Drug: Tenecteplase
- Control group (Other): standard stroke care based on national guideline
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — intravenous tenecteplase (0.25 mg/kg, a single bolus over 5 to 10 seconds, a maximum of 25 mg).

SUMMARY:
To date, the benefit of intravenous thrombolysis is confined within 4.5 hours of onset for acute ischemic stroke (AIS) patients without advanced neuroimaging selection. Unpublished pilot EXIT-BT (EXtending the tIme window of Thrombolysis by ButylphThalide up to 6 Hours after onset) suggest the safety, feasibility and potential benefit of intravenous tenecteplase (TNK) in AIS within 4.5 to 6 hours of onset. The current study aims to investigate the efficacy and safety of TNK for AIS within 4.5 to 6 hours of onset.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Acute ischemic stroke confirmed by non-contrast computed tomography and use of CTA for assessment of LVO as determined by local investigators;
* The time from last known well to treatment: 4.5 - 6 hours;
* NIHSS ≥ 4 at randomization;
* First stroke onset or past stroke without obvious neurological deficit (mRS≤1);
* Uncertainty over the benefits and risks of thrombolysis by researcher;
* Signed informed consent.

Exclusion Criteria:

* Pre-stroke disability (mRS≥2);
* Planned intravenous thrombolysis based on WAKE-UP or EXTEND study criterion;
* Any contraindication to intravenous thrombolysis: Obvious head injury or stroke within 3 months; Subarachnoid or intracranial hemorrhage; History of intracranial hemorrhage; Intracranial tumor, arteriovenous malformation or aneurysm; Intracranial or spinal cord surgery within 3 months; Myocardial infarction within 3 months; Major surgery within 1 month; Gastrointestinal or urinary tract hemorrhage within the previous 30 days; Arterial puncture at a noncompressible site within the previous seven days; Active internal hemorrhage; Coagulation abnormalities: platelet count of <100000/mm3; Aortic arch dissection; Heparin therapy within 24 hours; Infective endocarditis; Oral warfarin is being taken and INR>1.6 or APTT abnormal; Systolic pressure ≥185 mmHg or diastolic pressure ≥110 mmHg; Blood glucose < 50 mg/dl (2.7mmol/L); Neurological deficit after epileptic seizures;
* Pregnancy;
* Allergy to test drugs;
* Comorbidity with other serious diseases;
* Participating in other clinical trials within 3 months;
* Patients not suitable for the study considered by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
proportion of modified Rankin Scale (mRS) 0-1 | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome

SECONDARY OUTCOMES:
proportion of modified Rankin Scale (mRS) 0-2 | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
ordinal distribution of modified Rankin Scale (mRS) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
change in National Institute of Health stroke scale (NIHSS) score | 24 (-6/+12) hours
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
change in National Institute of Health stroke scale (NIHSS) score | 10±2 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
occurrence of early neurological improvement (ENI) | 24 (-6/+12) hours
  ENI is defined as more than 4-point decrease in National Institute of Health stroke scale score
new stroke or other vascular event(s) | 90±7 days
all-cause mortality | 90±7 days
symptomatic intracranial hemorrhage (sICH) | 24 (-6/+12) hours
  sICH is defined as parenchymal hematoma type 1 or 2 (PH1 or PH2), remote intraparenchymal hematoma (RIH), subarachnoid hemorrhage, or intraventricular hemorrhage on head CT/MRI scan causally associated with clinically significant neurological deterioration (NIHSS score ≥4 point increase) in the opinion of the clinical investigator or independent safety monitor.
intracranial hemorrhage | 24 (-6/+12) hours
  any evidence of bleeding on the head CT scan, classified by the Heidelberg Bleeding Classification
major systemic bleeding event | 24 (-6/+12) hours
any bleeding event | 24 (-6/+12) hours

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hui-Sheng Chen, Shenyang, None Selected
  - Department of Neurology, General Hospital of Northern Theater Command, Shenyang

IPD SHARING:
Plan to Share IPD: Undecided